CLINICAL TRIAL: NCT03626220
Title: Evaluation the Efficacy of Acupuncture in Chemotherapy Induced Peripheral Neuropathy
Brief Title: Acupuncture on Chemotherapy-induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chen Huang, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH106-REC2-117
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Randomized Controlled Trial; Breast Cancer; Chemotherapy-induced Peripheral Neuropathy; Acupuncture
Keywords: acupuncture; chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: 1. The acupuncture group: Acupuncture treatment will be performed for 9 weeks. The frequency of acupuncture will be twice a week for the first six weeks, and once a week for the following three weeks. 30 minutes needling at each treatment. Acupuncture points include Baihui(GV20), Qihai(CV6), Quchi(LI11), Hegu(LI4), Neiguan(P6), or Shenmen(HT7) for upper limbs. For plantar numbness, choose two acupoints to use in turn; use Weizhong(BL40), Sanyinjiao(SP6), or Zusanli(ST36) for lower limbs. If severe numbness occurred, Taixi(KI3) or Yongquan(K1) should be added for feet numbness. "De qi" sensation, such as soreness, numbness, pain, etc. will be achieved at each acupoints .
  2. The Controlled group: Acupuncture with superficial needling 0.5 cun (estimated 1cm with deviation depends on the body size of each participants) away from the acupoints, which only superficially penetrated the skin without feeling of "De Qi" sensation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The acupuncture group (Experimental): Acupuncture treatment will be performed for 9 weeks. Acupuncture treatment will be performed for 9 weeks. The frequency of acupuncture will be twice a week for the first six weeks, and once a week for the following three weeks. 30 minutes needling at each treatment. Acupuncture points include Baihui(GV20), Qihai(CV6), Quchi(LI11), Hegu(LI4), Neiguan(P6), or Shenmen(HT7) for upper limbs. For plantar numbness, choose two acupoints to use in turn; use Weizhong(BL40), Sanyinjiao(SP6), or Zusanli(ST36) for lower limbs. If severe numbness occurred, Taixi(KI3) or Yongquan(K1) should be added for feet numbness. "De qi" sensation, such as soreness, numbness, pain, etc. will be achieved at each acupoints .
  Interventions: Other: acupuncture
- The controlled group (Sham Comparator): Acupuncture with superficial needling 0.5 cun (estimated 1cm with deviation depends on the body size of each participants) away from the acupoints, which only superficially penetrated the skin without feeling of "De Qi" sensation.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — More than five years of experienced certified acupuncturists performed all treatments using the study protocol and administered to all participants. The acupoints selection principle was based on the Bi syndrome(the impediment disease) recorded in the Huangdi's Internal Classic, the Traditional Chinese medicine literature. Disposable sterile stainless steel needles (CASOON, Wuxi Jiajian Medical Instrument Company, Limited., Jiangsu, China) with 0.3mm in diameter and 40mm in length, were inserted into the prespecified acupoints

SUMMARY:
Peripheral neuropathy is currently the second most common side effect after chemotherapy, second only to the side effects of blood toxicity. A variety of chemotherapy drugs may induce peripheral neurotoxicity and cause by the cumulative dose of chemotherapy drugs. Symptoms include sensory paresthesia, feeling dullness or numbness, glove-like feeling distributed in the palm. The currently most effective way is to interrupt the treatment or adjust the dose of chemotherapeutic drugs, but it is easy to make patients discontinue chemotherapy. The purpose of this study is to explore the impact of acupuncture on neurological symptoms and quality of life. Three kinds of questionnaires will be used:(1) Brief pain inventory- short form to assess the extent of pain, and the impact of daily life. (2) the Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group- Neurotoxicity(FACT/GOG-NTX)-13 (Version 4) to assess changes in neurological symptoms; (3) World Health Organization Quality of Life Scale-(WHOQOL-BREF) to assess changes in the quality of life of patients. The course of treatment was evaluated for nine weeks. Changes in neurological function and quality of life will be evaluated before treatment, the third week of treatment, the sixth week of treatment, till the ninth week. The aim of this study is to confirm that acupuncture can improve peripheral neuropathy after chemotherapy, in order to enhance breast cancer patients' quality of life, and provide the new opportunity for integrative therapy between Chinese and Western medicine.

Keywords：acupuncture , chemotherapy-induced peripheral neuropathy

DETAILED DESCRIPTION:
(I) Background of the research A variety of neurotoxic chemotherapeutic agents, including platinums (e.g. cisplatin, carboplatin, and oxaliplatin), taxanes (e.g. paclitaxel and docetaxel), and vinca alkaloids (e.g. vincristine and vinblastine), thalidomide and bortezomib, may induce peripheral neuropathy. Generally speaking, sensory nerve dysfunction is more common than motor involvement. It causes hands and feet to feel tingling, dullness or numbness symmetrically, which will be a glove-like ("glove-and-stocking type") sensation distributed in palms and soles. Patient's touch, vibration, and proprioception senses may be impaired under clinical examinations.

chemotherapy-induced peripheral neuropathy(CIPN) relates to the cumulative doses of chemotherapeutic agents. Sometimes, when chemotherapy is stopped, neuropathy symptoms may continue or worsen, which is called a "costing phenomenon". Nerve damaging usually starts from ends of the extremities, while individual doses were accumulated, it gradually extends to proximal joints or ganglions. CIPN is currently the second most common side, next to hematotoxicity. Within thirty days after chemotherapy, 68.1% of patients may develop CIPN, most of which can be relieved or improved, but there are still 30-83% symptoms persist over 6 months.

At present, the most effective way to treat CIPN is to stop the treatment protocol or adjust doses of chemotherapy; however, it affects the effect of chemotherapy in degrading tumor growth. Plenty of pharmacological or non-pharmacological treatments are still under investigation, such as antioxidant medication (e.g. Acetyl-L-carnitine, glutamine, vit B12, fish oil, etc.), anxiolytics (e.g. venlafaxine), neuroprotective agents (e.g. infusion of calcium ions, magnesium ions), food supplements, acupuncture, light stimulation, etc. Acupuncture with the advantages of clinically effective, easy-practice and relatively safe, few studies revealed its effect on CIPN, however, there is still a lack of large clinical trials to evaluate its effectiveness.

(ii) Purpose of the research To investigate the efficacy of acupuncture on peripheral neuropathy after chemotherapy administration in patients with breast cancer.

(iii) Importance of the research Current studies revealed that acupuncture might be effective on CIPN, however, insufficient number of participants or lack of control groups limit the quality of clinical studies. Therefore, the aim of our study to conduct a randomized controlled clinical trial to evaluate the efficacy of acupuncture on peripheral neuropathy caused by chemotherapy.

ELIGIBILITY:
The inclusion criteria will be: female more than 20 years of age; breast cancer with early stage at I-III; had completed chemotherapy; the neurotoxic chemotherapeutic agents included taxanes, platinums, or others; less than grade three in the Eastern Cooperative Oncology Group (ECOG) status; higher than grade one in National Cancer Institute-common terminology criteria for adverse events(NCI-CTCAE) scale.

The exclusion criteria will be: having less than three months in mean survival time, history of diabetic neuropathy before chemotherapy administration, history of other preexisting peripheral neuropathy, other inflammatory or metabolic arthritis, severe blood coagulation diseases or with latent bleeding tendency, unstable cardiovascular diseases, or other preexisting muscle-skeletal diseases.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chen Huang, M.S., Principal Investigator — An Nan Hospital, China Medical University, Tainan, Taiwan, R.O.C.
Locations (1):
- An Nan Hospital, China Medical University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franconi G, Manni L, Schroder S, Marchetti P, Robinson N. A systematic review of experimental and clinical acupuncture in chemotherapy-induced peripheral neuropathy. Evid Based Complement Alternat Med. 2013;2013:516916. doi: 10.1155/2013/516916. Epub 2013 Jul 24. PMID 23983788
- [Background] Park SB, Goldstein D, Krishnan AV, Lin CS, Friedlander ML, Cassidy J, Koltzenburg M, Kiernan MC. Chemotherapy-induced peripheral neurotoxicity: a critical analysis. CA Cancer J Clin. 2013 Nov-Dec;63(6):419-37. doi: 10.3322/caac.21204. PMID 24590861
- [Result] Greenlee H, Crew KD, Capodice J, Awad D, Buono D, Shi Z, Jeffres A, Wyse S, Whitman W, Trivedi MS, Kalinsky K, Hershman DL. Randomized sham-controlled pilot trial of weekly electro-acupuncture for the prevention of taxane-induced peripheral neuropathy in women with early stage breast cancer. Breast Cancer Res Treat. 2016 Apr;156(3):453-464. doi: 10.1007/s10549-016-3759-2. Epub 2016 Mar 25. PMID 27013473
- [Result] Wong R, Major P, Sagar S. Phase 2 Study of Acupuncture-Like Transcutaneous Nerve Stimulation for Chemotherapy-Induced Peripheral Neuropathy. Integr Cancer Ther. 2016 Jun;15(2):153-64. doi: 10.1177/1534735415627926. Epub 2016 Apr 29. PMID 27130723
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/27013473
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/27130723
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/23983788
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/24590861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 269 patients diagnosed with breast cancer were screened from June 2018 to July 2020. Of 61 potentially eligible patients, 20 (32.8%) were enrolled and randomized as 10 in the acupuncture group and 10 in the sham acupuncture group. 208 ineligible patients were excluded, and 41 patients declined to participate in our study.
Groups:
- The Acupuncture Group: Acupuncture treatment will be performed for 9 weeks. The frequency of acupuncture will be twice a week for the first six weeks, and once a week for the following three weeks. 30 minutes needling at each treatment. Acupuncture points include Baihui(GV20), Qihai(CV6), Quchi(LI11), Hegu(LI4), Neiguan(P6), and Shenmen(HT7) for upper limbs. For palm numbness, choose two acupoints to use in turn; use Weizhong(BL40), Sanyinjiao(SP6), and Zusanli(ST36) for lower limbs. For the acupuncture points, Taixi(KI3) and Yongquan(K1) should be added for foot numbness. "De qi" sensation, such as soreness, numbness, pain, etc. will be achieved at each acupoints .
  acupuncture: More than five years of experienced certified acupuncturists performed all treatments using the study protocol and administered to all participants. The acupoints selection principle was based on the Bi syndrome(the impediment disease) recorded in the Huangdi's Internal Classic, the Traditional Chinese medicine literature. Disposable sterile stainless steel needles (CASOON, Wuxi Jiajian Medical Instrument Company, LTD., Jiangsu, China) with 0.3mm in diameter and 40mm in length, were inserted into the prespecified acupoints
- The Controlled Group: Acupuncture with superficial needling 0.5 cun (estimated 1cm with deviation depends on the body size of each participants) away from the acupoints, which only superficially penetrated the skin without feeling of "De Qi" sensation.
  acupuncture: More than five years of experienced certified acupuncturists performed all treatments using the study protocol and administered to all participants. The acupoints selection principle was based on the Bi syndrome(the impediment disease) recorded in the Huangdi's Internal Classic, the Traditional Chinese medicine literature. Disposable sterile stainless steel needles (CASOON, Wuxi Jiajian Medical Instrument Company, Limited, Jiangsu, China) with 0.3mm in diameter and 40mm in length, were inserted into the prespecified acupoints
Period: Overall Study
Arm/Group | The Acupuncture Group | The Controlled Group
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- The Controlled Group: Acupuncture with superficial needling 0.5 cun (estimated 1cm with deviation depends on the body size of each participants) away from the acupoints, which only superficially penetrated the skin without feeling of "De Qi" sensation.
  acupuncture: More than five years of experienced certified acupuncturists performed all treatments using the study protocol and administered to all participants. The acupoints selection principle was based on the Bi syndrome(the impediment disease) recorded in the Huangdi's Internal Classic, the Traditional Chinese medicine literature. Disposable sterile stainless steel needles (CASOON, Wuxi Jiajian Medical Instrument Company, LTD., Jiangsu, China) with 0.3mm in diameter and 40mm in length, were inserted into the prespecified acupoints
- Total: Total of all reporting groups
Arm/Group | The Acupuncture Group | The Controlled Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.10 (11.07) | 52.10 (11.18) | 49.60 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 10 | 10 | 20
Eastern Cooperative Group(ECOG) performance status [Count of Participants; unit: Participants] — Grade: ECOG performance status 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    Grade 0 | 10 | 9 | 19
    Grade 1 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Average Pain Severity in the Brief Pain Inventory-Short Form(BPI-SF)
Description: The average pain severity was chosen as the primary assessment as neuropathy symptoms based on its ability to detect neuropathic pain in cancer patients, as well as its use to assess CIPN symptoms in other controlled clinical trials.The BPI-SF assesses pain when responding to the questionnaire (right now) and at its worst, least, and average pain severity in the last 24 h. The items range from 0 to 10 (0 = no pain; 10 = worst pain). The higher the pain severity scores, the worse the degree of pain experienced by the patient. We analyzed the data (1) within group analysis: compared the data at week 6 with baseline, and the data at week 9 with baseline from each group. (2) between group analysis: compared the acupuncture group and sham acupuncture group at week 6 and week 9. (3) the between group differences of the changes from week 6 to baseline and from week 9 to baseline.
Time Frame: We measured the average pain severity 4 times within 9 weeks [at baseline (before the first treatment) and week 3, week 6, and week 9 during the protocol].
Population: * In the acupuncture group, one subject withdrew from the trial because of needle phobia after the third week of treatment, and another subject withdrew from the trial because of cellulitis in the radiation treatment site after completing the sixth week of treatment
  * In the placebo group, one subject did not record the scoring result after completing the sixth week of acupuncture treatment because of the omission to fill in this scale
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- The Acupuncture Group: Acupuncture treatment will be performed for 9 weeks. The frequency of acupuncture will be twice a week for the first six weeks, and once a week for the following three weeks. 30 minutes needling at each treatment. Acupuncture points include Baihui(GV20), Qihai(CV6), Quchi(LI11), Hegu(LI4), Neiguan(P6), or Shenmen(HT7) for upper limbs. For plantar numbness, choose two acupoints to use in turn; use Weizhong(BL40), Sanyinjiao(SP6), or Zusanli(ST36) for lower limbs. If severe numbness occurred, Taixi(KI3) or Yongquan(K1) should be added for feet numbness. "De qi" sensation, such as soreness, numbness, pain, etc. will be achieved at each acupoints .
Arm/Group | The Acupuncture Group | The Controlled Group
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 3.10 (2.33) | 3.10 (1.79)
  Week 3: number analyzed (Participants) | 9 | 10
  Week 3 | 1.72 (1.48) | 3.50 (2.27)
  Week 6: number analyzed (Participants) | 8 | 9
  Week 6 | 1.63 (0.92) | 2.78 (2.82)
  Week 9: number analyzed (Participants) | 8 | 10
  Week 9 | 0.88 (1.13) | 2.70 (2.00)
  Changes at week 6: number analyzed (Participants) | 8 | 9
  Changes at week 6 | -1.63 (1.85) | -0.11 (2.71)
  Changes at week 9: number analyzed (Participants) | 8 | 10
  Changes at week 9 | -2.38 (2.39) | -0.40 (2.07)

2. Secondary Outcome: Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group- Neurotoxicity(FACT/GOG-NTX)-13
Description: The 27-item FACT-G evaluated the quality of life of patients undergoing cancer therapy over the past 7 days. The question is rated on a five-point scale, from 0 to 4 (0= not at all; 4= very much) and summed ( total score range= 0-108). An increase in scores represents an improvement in the overall quality of life.The 13-item Ntx subscale measures the severity and impact of neurotoxicity symptoms over the past seven days. Items are rated on a five-point scale, scored from 0 to 4 and summed ( total score range= 0-52). Higher scores on the neurotoxicity scale indicate improvements in neurotoxic symptoms.
  The 40-item FACT/GOG-Ntx total score represents the sum of the FACT-G and Ntx subscale (total score range=0-160).The FACT/GOG-Ntx trial outcome index (TOI) contained the scores of the PWB, FWB, and FACT/GOG-Ntx subscale (total score range= 0-104).We analyzed the data (1) within group analysis(2) between group analysis(3) the changes between group analysis
Time Frame: 4 times within 9 weeks: at baseline (before the first treatment) and week 3, week 6, and week 9 during the protocol
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Acupuncture Group | The Controlled Group
Number analyzed (Participants) | 10 | 10
score on a scale
  NtxS-baseline | 37.60 (6.08) | 33.90 (7.87)
  NtxS-week 3: number analyzed (Participants) | 9 | 10
  NtxS-week 3 | 37.89 (6.01) | 33.62 (6.52)
  NtxS-week 6: number analyzed (Participants) | 8 | 9
  NtxS-week 6 | 41.00 (6.72) | 36.44 (8.71)
  NtxS-week 9: number analyzed (Participants) | 8 | 10
  NtxS-week 9 | 40.88 (7.72) | 35.90 (5.92)
  NtxS-Changes at week 6: number analyzed (Participants) | 8 | 9
  NtxS-Changes at week 6 | 3.63 (5.07) | 1.56 (7.55)
  NtxS-Changes at wee 9: number analyzed (Participants) | 8 | 10
  NtxS-Changes at wee 9 | 3.50 (4.90) | 2.00 (6.96)
  TOI-baseline | 76.60 (14.74) | 67.80 (15.25)
  TOI-week 3: number analyzed (Participants) | 9 | 10
  TOI-week 3 | 77.04 (16.03) | 69.57 (13.39)
  TOI-week 6: number analyzed (Participants) | 8 | 9
  TOI-week 6 | 81.75 (19.03) | 73.44 (16.54)
  TOI-week 9: number analyzed (Participants) | 8 | 10
  TOI-week 9 | 80.42 (20.58) | 74.60 (11.91)
  TOI-changes at week 6: number analyzed (Participants) | 8 | 9
  TOI-changes at week 6 | 6.63 (7.41) | 3.00 (14.34)
  TOI-changes at week 9: number analyzed (Participants) | 8 | 10
  TOI-changes at week 9 | 5.29 (6.31) | 6.80 (12.62)
  FACT-G score-baseline | 79.70 (16.35) | 69.73 (14.19)
  FACT-G score-week 3: number analyzed (Participants) | 9 | 10
  FACT-G score-week 3 | 77.96 (20.02) | 73.20 (15.95)
  FACT-G score-week 6: number analyzed (Participants) | 8 | 9
  FACT-G score-week 6 | 80.08 (19.80) | 73.49 (16.16)
  FACT-G score-week 9: number analyzed (Participants) | 8 | 10
  FACT-G score-week 9 | 77.54 (21.55) | 77.73 (11.10)
  FACT-G score-changes at week 6: number analyzed (Participants) | 8 | 9
  FACT-G score-changes at week 6 | 1.06 (2.89) | 1.66 (12.94)
  FACT-G score-changes at week 9: number analyzed (Participants) | 8 | 10
  FACT-G score-changes at week 9 | -1.48 (5.51) | 8 (10.31)
  FACT/GOG-Ntx total score-baseline | 117.30 (20.56) | 103.63 (19.75)
  FACT/GOG-Ntx total score-week 3: number analyzed (Participants) | 9 | 10
  FACT/GOG-Ntx total score-week 3 | 115.85 (23.80) | 106.82 (18.34)
  FACT/GOG-Ntx total score-week 6: number analyzed (Participants) | 8 | 9
  FACT/GOG-Ntx total score-week 6 | 121.08 (25.93) | 109.93 (20.79)
  FACT/GOG-Ntx total score-week 9: number analyzed (Participants) | 8 | 10
  FACT/GOG-Ntx total score-week 9 | 118.42 (28.55) | 113.43 (12.80)
  FACT/GOG-Ntx total score-changes at week 6: number analyzed (Participants) | 8 | 9
  FACT/GOG-Ntx total score-changes at week 6 | 4.69 (7.39) | 3.21 (18.40)
  FACT/GOG-Ntx total score-changes at week 9: number analyzed (Participants) | 8 | 10
  FACT/GOG-Ntx total score-changes at week 9 | 2.02 (8.01) | 9.80 (14.30)

3. Secondary Outcome: World Health Organization Quality of Life Scale(WHOQOL)-BREF (Taiwan Version)
Description: WHOQOL-BREF Taiwan version was validated to be a good clinical tool across five kinds of Taiwanese cancer survivors. There are a total 28 items by adding 2 additional items to account for Taiwanese cultural adaptations. Item scores range from 1 to 5 (1 =the worst condition; 5=the best condition), except for 3 items (Ph1, Ph2, and Ps6), which are reverse coded. Each domain in the scale can be translated into two ranges of domain scores (0-100 and 4-20), and we used 0-100 scale in this study. The Higher scores in each domain indicate the better quality of life for patients with cancers We analyzed the data (1) within group analysis: compared post-treatment with baseline. (2) between group analysis: compared the acupuncture group and sham acupuncture group at week 9. (3) the between group differences of the changes from post-treatment to baseline.
Time Frame: We measured 2 times within 9 weeks: before and after treatment
Population: - In the acupuncture group, one subject withdrew from the trial because of needle phobia after the third week of treatment, and another subject withdrew from the trial because of cellulitis in the radiation treatment site after completing the sixth week of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- The Acupuncture Group: : Acupuncture treatment will be performed for 9 weeks. The frequency of acupuncture will be twice a week for the first six weeks, and once a week for the following three weeks. 30 minutes needling at each treatment. Acupuncture points include Baihui(GV20), Qihai(CV6), Quchi(LI11), Hegu(LI4), Neiguan(P6), or Shenmen(HT7) for upper limbs. For plantar numbness, choose two acupoints to use in turn; use Weizhong(BL40), Sanyinjiao(SP6), or Zusanli(ST36) for lower limbs. If severe numbness occurred, Taixi(KI3) or Yongquan(K1) should be added for feet numbness. "De qi" sensation, such as soreness, numbness, pain, etc. will be achieved at each acupoints .
Arm/Group | The Acupuncture Group | The Controlled Group
Number analyzed (Participants) | 10 | 10
score on a scale
  Physical health-baseline | 60.80 (15.97) | 55.20 (12.69)
  Physical health-post-Tx: number analyzed (Participants) | 8 | 10
  Physical health-post-Tx | 60.88 (17.88) | 59.50 (11.34)
  Physical health-Changes at post-Tx: number analyzed (Participants) | 8 | 10
  Physical health-Changes at post-Tx | 3.63 (13.52) | 4.30 (13.36)
  Psychological-baseline | 51.40 (13.79) | 45.20 (16.58)
  Psychological-post-Tx: number analyzed (Participants) | 8 | 10
  Psychological-post-Tx | 55.50 (18.62) | 52.50 (13.52)
  Psychological-changes at post-Tx: number analyzed (Participants) | 8 | 10
  Psychological-changes at post-Tx | 6.13 (11.79) | 7.30 (8.14)
  Social relationships-baseline | 62.10 (9.56) | 54.50 (10.22)
  Social relationships-post Tx: number analyzed (Participants) | 8 | 10
  Social relationships-post Tx | 68.00 (11.15) | 58.90 (10.80)
  Social relationships-changes at post-Tx: number analyzed (Participants) | 8 | 10
  Social relationships-changes at post-Tx | 6.88 (9.69) | 4.40 (11.90)
  Environment-baseline | 61.90 (8.20) | 61.40 (13.02)
  Environment-post Tx: number analyzed (Participants) | 8 | 10
  Environment-post Tx | 61.75 (10.33) | 66.30 (11.84)
  Environment-changes at post-Tx: number analyzed (Participants) | 8 | 10
  Environment-changes at post-Tx | -1.63 (11.60) | 4.90 (10.97)

4. Secondary Outcome: Touch Test Sensory Evaluator
Description: Measurements were performed using a set of 20 von Frey monofilaments(Semmes-Weinstein Von Frey Aesthesiometer, Stoelting Co. 620 Wheat Lane, Wood Dale, IL, U.S.A.), with evaluator size/target forces from 1.65/0.008 gto 6.65/300 g. Each monofilament was calibrated to a target force in grams (g) within a 5% standard deviation. Thresholds for categories of tactile perception were defined by the filament manufacturer as follows: normal ; diminished light touch; diminished protective sensation; loss of protective sensation; deep pressure sensation only . All tests were performed by an independent assessor who was unaware of the allocation of randomization. All the procedures followed the operation manual provided by the filament manufacturer. Measuring sites include: LHT(Left hand's middle fingertip);LHP(Left hand's palm);RHT(Right hand's middle fingertip);RHP(Right hand's palm);LFT(Left foot's big toe tip);LFP(Left foot's plantar);RFT(Right foot's big toe tip);RFP(Right foot's plantar)
Time Frame: 2 times within 9 weeks: before and after treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | The Acupuncture Group | The Controlled Group
Number analyzed (Participants) | 10 | 10
grams
  LHT-baseline | 1.64 (1.87) | 1.62 (1.41)
  LHT-post-Tx: number analyzed (Participants) | 8 | 10
  LHT-post-Tx | 0.41 (0.66) | 1.82 (2.28)
  LHT-changes at post-Tx: number analyzed (Participants) | 8 | 10
  LHT-changes at post-Tx | -1.54 (2.12) | 0.20 (2.51)
  LHP-baseline | 2.60 (4.69) | 1.98 (2.89)
  LHP-post-Tx: number analyzed (Participants) | 8 | 10
  LHP-post-Tx | 0.25 (0.23) | 1.44 (1.99)
  LHP-changes at post-Tx: number analyzed (Participants) | 8 | 10
  LHP-changes at post-Tx | -2.92 (5.20) | -0.54 (1.73)
  RHT-baseline | 1.52 (1.35) | 1.74 (1.31)
  RHT-post-Tx: number analyzed (Participants) | 8 | 10
  RHT-post-Tx | 0.37 (0.29) | 1.25 (1.78)
  RHT-changes at post-Tx: number analyzed (Participants) | 8 | 10
  RHT-changes at post-Tx | -1.43 (1.37) | -0.50 (2.20)
  RHP-baseline | 2.50 (4.53) | 1.91 (1.85)
  RHP-post-Tx: number analyzed (Participants) | 8 | 10
  RHP-post-Tx | 0.28 (0.20) | 1.27 (1.77)
  RHP-changes at post-Tx: number analyzed (Participants) | 8 | 10
  RHP-changes at post-Tx | -2.75 (5.06) | -0.64 (1.13)
  LFT-baseline | 14.02 (30.57) | 10.30 (17.99)
  LFT-post-Tx: number analyzed (Participants) | 8 | 10
  LFT-post-Tx | 2.50 (2.49) | 3.50 (3.41)
  LFT-changes at post-Tx: number analyzed (Participants) | 8 | 10
  LFT-changes at post-Tx | -14.87 (34.46) | -6.80 (16.04)
  LFP-baseline | 20.66 (56.17) | 9.61 (18.09)
  LFP-post-Tx: number analyzed (Participants) | 8 | 10
  LFP-post-Tx | 2.35 (5.13) | 3.24 (4.60)
  LFP-changes at post-Tx: number analyzed (Participants) | 8 | 10
  LFP-changes at post-Tx | -23.40 (57.43) | -6.36 (13.99)
  RFT-baseline | 12.80 (17.30) | 5.28 (7.55)
  RFT-post-Tx: number analyzed (Participants) | 8 | 10
  RFT-post-Tx | 2.43 (2.94) | 4.94 (4.71)
  RFT-changes at post-Tx: number analyzed (Participants) | 8 | 10
  RFT-changes at post-Tx | -12.45 (19.99) | -0.34 (7.15)
  RFP-baseline | 6.46 (6.53) | 9.36 (18.01)
  RFP-post-Tx: number analyzed (Participants) | 8 | 10
  RFP-post-Tx | 2.87 (5.06) | 3.94 (3.77)
  RFP-changes at post-Tx: number analyzed (Participants) | 8 | 10
  RFP-changes at post-Tx | -4.93 (6.11) | -5.41 (15.95)

5. Other Pre Specified Outcome: Explore the Neuroprotective Mechanism of Acupuncture
Description: 15 cc of blood samples will be drawn before and after 15 sessions of treatments from participants in both groups. The blood samples will be analyzed by enzyme-linked immunosorbent assay (ELISA) for tumor necrosis factor-alfa and interleukin- 6, interleukin-10 and brain-derived nuerotrophic factor to evaluate the differences in the inflammation state of peripheral nervous system within and between groups.
Time Frame: 2 times within 9 weeks: before and after treatment
Population: Due to the difficulty of the execution in the hospital, the execution was abandoned
Arm/Group | The Acupuncture Group | The Controlled Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: A total of nine weeks from the start of the study to the end of the study
Arm/Group | The Acupuncture Group | The Controlled Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03626220/Prot_SAP_000.pdf